CLINICAL TRIAL: NCT03628079
Title: A Phase 2a TDM-guided Clinical Study on the Safety and Efficacy of Mebendazole in Patients With Advanced Gastrointestinal Cancer or Cancer of Unknown Origin
Brief Title: A Clinical Safety and Efficacy Study of Mebendazole on GI Cancer or Cancer of Unknown Origin.
Acronym: RepoMeb
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of effect
Sponsor: Repos Pharma (Industry)
Collaborators: Uppsala University (Other); Uppsala University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP-2017-001
Record Dates: First submitted 2018-06-17; First posted 2018-08-14 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Cancer of the Gastrointestinal Tract; Cancer of Unknown Origin
MeSH Terms: conditions — Gastrointestinal Neoplasms; Neoplasms, Unknown Primary | interventions — Mebendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study (Experimental): ReposMBZ 100 mg capsule by mouth followed by 8h PK sampling to decide the initial daily dose.
  Treatment: Repos MBZ capsules by mouth twice daily for 16 weeks, daily dose 50mg-4g, based on the serum level of mebendazole.
  Interventions: Drug: ReposMBZ

INTERVENTIONS:
Drug: ReposMBZ — Capsules 50mg, 100mg, 200mg
  Other Names: Mebendazole

SUMMARY:
This study will evaluate the safety and efficacy of mebendazole (ReposMBZ) in patient with advanced gastrointestinal cancer or cancer of unknown origin. All patients will be given ReposMBZ for 16 weeks continuous treatment, individually dosed based on the serum concentration of mebendazole.

DETAILED DESCRIPTION:
Mebendazole has been used extensively during long time for local gut helminthic infections at low dose but also at considerably higher doses during months to years against invasive echinococcus infections. Recent research has now clearly indicated that mebendazole has anticancer effect. Given these observations and the experience of excellent tolerance to mebendazole the current clinical trial protocol is based on the repositioning strategy to more extensively investigate whether mebendazole could be developed into a useful anticancer drug.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Histologically confirmed diagnosis of squamous cell cancer or adenocarcinoma, including primary cancer of the liver, of the gastrointestinal tract or cancer of unknown origin.
3. Measurable disease according to RECIST 1.1.
4. Defined time to tumour progression on the standard/experimental treatment preceding the trial treatment.
5. Locally advanced or metastatic disease not amenable to standard treatment, i.e. progress on standard therapy or observed/expected intolerance to standard therapy.
6. - (removed via Amendment 1)
7. Pharmacological treatment attempt considered reasonable.
8. Females of childbearing potential should use adequate contraception throughout the study;

   1. Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal)
   2. Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable)
   3. Intrauterine device (IUD)
   4. Intrauterine hormone-releasing system (IUS)
   5. Bilateral tubal occlusion
   6. Vasectomized partner
   7. Sexual abstinence
9. Signed informed consent.

Exclusion Criteria:

1. Anti-tumour therapy within 3 weeks prior to study drug administration day
2. Ongoing infection or other major recent or ongoing disease that, according to the investigator, poses an unacceptable risk to the patient.
3. WHO performance status ≥ 2.
4. Child-Pugh B or C liver function status if hepatocellular carcinoma.
5. Inadequate laboratory parameters reflecting major organ function i.e.:

   1. neutrophils ≤ 1,3 x 109/l
   2. platelets ≤ 100 x 109/l
   3. bilirubin > 1.5 x upper limit of normal (ULN)
   4. Alanine aminotransferase (ALAT) > 5 x ULN
   5. Glomerular filtration rate (GFR) <50 ml/min (calculated from P-creatinine)
   6. Prothrombin complex/INR outside normal range
6. Current active participation in any other interventional clinical study.
7. Contraindications to the investigational product, e.g. known or suspected hypersensitivity or inability to oral drug administration.
8. Pregnancy or lactation.
9. Lack of suitability for participation in the study, e g expected difficulties to follow the protocol procedures, as judged by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) probably or possibly related to ReposMBZ | From date of first dose, up to 30 days after last dose of ReposMBZ or start of new treatment, whatever comes first, assessed up to 20 weeks after start of treatment phase.
  AEs graded according to CTCAE 4.03.
Changes in plasma Albumin over time | From date of first dose, up to 30 days after last dose of ReposMBZ or start of new treatment, whatever comes first, assessed up to 20 weeks after start of treatment phase.
  Blood Chemistry (plasma): Albumin (g/L)
Changes in C-reactive protein (CRP) over time | From date of first dose, up to 30 days after last dose of ReposMBZ or start of new treatment, whatever comes first, assessed up to 20 weeks after start of treatment phase.
  Blood chemistry (plasma): CRP (mg/L)
Changes in plasma Sodium, Potassium, Calcium and Glucose over time | From date of first dose, up to 30 days after last dose of ReposMBZ or start of new treatment, whatever comes first, assessed up to 20 weeks after start of treatment phase.
  Blood chemistry (plasma): Sodium, Potassium, Calcium, Glucose (mmol/L)
Changes in plasma Bilirubin over time | From date of first dose, up to 30 days after last dose of ReposMBZ or start of new treatment, whatever comes first, assessed up to 20 weeks after start of treatment phase.
  Blood chemistry (plasma): Bilirubin (µmol/L)
Changes in plasma ALAT (alanine aminotransferase), ASAT (aspartate aminotransferase), LDH (lactate dehydrogenase), ALP (alkaline phosphatase) over time | From date of first dose, up to 30 days after last dose of ReposMBZ or start of new treatment, whatever comes first, assessed up to 20 weeks after start of treatment phase.
  Blood chemistry (plasma): ALAT, ASAT, LDH, ALP (µkat/L)
Changes in Haemoglobin over time | From date of first dose, up to 30 days after last dose of ReposMBZ or start of new treatment, whatever comes first, assessed up to 20 weeks after start of treatment phase.
  Haematology: Haemoglobin (g/L)
Changes in red, white and platelet blood cell count over time | From date of first dose, up to 30 days after last dose of ReposMBZ or start of new treatment, whatever comes first, assessed up to 20 weeks after start of treatment phase.
  Haematology: RBC (red blood cell count), White blood cells with differential count and platelets (absolute count/L)
Changes in Activated Partial Thromboplastin Time (APTT) over time | From date of first dose, up to 30 days after last dose of ReposMBZ or start of new treatment, whatever comes first, assessed up to 20 weeks after start of treatment phase.
  Coagulation (plasma): APTT (s)
Changes in Prothrombin complex (PK/INR) over time | From date of first dose, up to 30 days after last dose of ReposMBZ or start of new treatment, whatever comes first, assessed up to 20 weeks after start of treatment phase.
  Coagulation (plasma): Prothrombin complex (INR)
Changes in blood pressure over time | From date of first dose, up to 30 days after last dose of ReposMBZ or start of new treatment, whatever comes first, assessed up to 20 weeks after start of treatment phase.
  Systolic and diastolic blood pressure (mmHg) Weight (kg)
Changes in heart rate over time | From date of first dose, up to 30 days after last dose of ReposMBZ or start of new treatment, whatever comes first, assessed up to 20 weeks after start of treatment phase.
  Supine heart rate (beats per minute)
Changes in body temperature over time. | From date of first dose, up to 30 days after last dose of ReposMBZ or start of new treatment, whatever comes first, assessed up to 20 weeks after start of treatment phase.
  Body temperature (Celsius degrees)
Tumour response: CT/MRI assessed according to RECIST 1.1 | From date of first dose ReposMBZ until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 24 months (end of study).
  Best overall radiological response Time to tumour progression (TTP) compared with TTP on the treatment just preceding this protocol.

SECONDARY OUTCOMES:
The peak serum concentration (Cmax) of ReposMBZ after single dose administration. | Pre-dose, 30 minutes, 60 minutes, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours.
  Cmax will be used to decide the starting dose in the treatment phase.
Area under the serum concentration versus time curve (AUC) for ReposMBZ | Pre-dose, 30 minutes, 60 minutes, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours.
  Analysis of serum concentration after single dose administration of ReposMBZ.
The Cmax serum concentration of ReposMBZ after repeated dose administration. | Pre-dose, 30 minutes, 60 minutes, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours (only up to the time point for Cmax after single dose), assessed up to 16 weeks after start of treatment phase.
  Cmax will be used to adjust the dose until target S-mebendazole level is reached and to show the individual variation of S-mebendazole concentration over time
Target S-mebendazole concentration after repeated dose administration. | From first dose in treatment phase and assessed up to 16 weeks after start of treatment phase.
  Number of patients that reach the steady state S-mebendazole target concentration.
Time to reach the steady state S-mebendazole target concentration after repeated dose administration.. | From first dose in treatment phase and assessed up to 16 weeks after start of treatment phase.
  Time from first dose in treatment phase until target S-mebendazole concentration is reached
Systemic immune activation. | From baseline up to 20 weeks after start of treatment phase, assessed up to 24 months (end of study).
  Change of cytokine levels in blood, evaluated by cytokine array.
Immune cell activation. | From baseline and up to 20 weeks after start of treatment phase, assessed up to 24 months (end of study).
  Up-regulation of activation markers compared to baseline, evaluated by flow cytometry.
Overall survival. | From date of first dose ReposMBZ to date of death, assessed up to 24 months (end of study).
  Months of survival from first dose until death of any cause.
Change in tumour load and TTP according to irRECIST | From date of first dose ReposMBZ until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 24 months (end of study).
  Best over all radiological response according to irRECIST 1.1.

OTHER OUTCOMES:
Association between ReposMBZ efficacy and properties of the diagnostic tumour tissue (optional) | Assessed up to 24 months (end of study).
  Genetic changes and infiltration of immune cells, grade, molecular subtype, gene and protein expression and tumour infiltration and subtypes of macrophages and lymphocytes.
Comparison of diagnostic tissue and a fresh tumour biopsy after 4 weeks of treatment at the target S-mebendazole concentration (optional). | Collected up to 20 weeks after start of treatment phase, assessed up to 24 months (end of study).
  Changes in the properties analysed in the archived tissue (baseline) and the fresh biopsy.
Association between S-mebendazole and efficacy and safety | From date of first dose until date of first documented progression or date of death, whichever comes fist, assessed up to 24 months (end of study).
  Mean S-mebendazole concentration during treatment phase in relation to safety (CTCAE 4.03 grade 3 and 4 toxicity) and efficacy (tumour response and TTP) respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of oncology, University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No